CLINICAL TRIAL: NCT03095001
Title: Chinese PLA Generation Hospital
Brief Title: Intraperitoneal Chemotherapy Alone or in Combination With Bevacizumab for Ovarian Cancer With Peritoneal Adhesion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, DuNan, Director of oncology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intraperitoneal bev
Record Dates: First submitted 2017-03-16; First posted 2017-03-29 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Peritoneal Adhesion
Keywords: bevacizumab; Intraperitoneal administration; Ovarian Cancer; Peritoneal Adhesion
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intraperitoneal bevacizumab+ carboplatin (Experimental): Intraperitoneal administration: intraperitoneal bevacizumab plus carboplatin every 3 weeks for 4-6 cycles
  Systemic chemotherapy: paclitaxel, iv. every 3 weeks for 4-6 cycles
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: paclitaxel
- Intraperitoneal carboplatin (Active Comparator): Intraperitoneal administration: intraperitoneal carboplatin every 3 weeks
  Systemic chemotherapy: paclitaxel, iv. every 3 weeks for 4-6 cycles
  Interventions: Drug: Carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 5mg/kg intraperitoneal administration every 3 weeks for 4-6 cycles
  Other Names: Avastin
  Arms: Intraperitoneal bevacizumab+ carboplatin
Drug: Carboplatin — carboplatin AUC=5 intraperitoneal administration every 3 weeks 4-6 cycles
Drug: paclitaxel — paclitaxel 175mg/m2, iv d1, every 3 weeks for 4-6 cycles

SUMMARY:
Background: Malignant peritoneal adhesion is a common complication and prognostic factor of ovarian cancer and other primary abdominal tumors. The incidence of peritoneal adhesion in advanced primary peritoneal tumor is 32-56%, which has increased by more than 10 times in the recent decade. Malignant peritoneal adhesion is closely associated with the morbidity and mortality of malignant intestinal obstruction. The peritoneal adhesion may aggravates the abdominal symptoms and reduce quality of life. Further, the peritoneal adhesion may impede treatment of primary tumor, such as operation or chemotherapy, lead to a poor prognosis.

Objective: This study aims to treat malignant peritoneal adhesion with the combination of antiangiogenic agent and chemotherapy, evaluate the efficacy and safety of intraperitoneal antiangiogenic agent plus chemotherapy. As explosive endpoints, we will examination the expression of VEGF-A in peritoneal cavity during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically and radiologically confirmed stage IV or postoperative recurrence ovarian cancer.
2. Age of 18-70, Karnofsky score higher than 80.
3. No severe functional damage of major organ, normal liver and kidney function.
4. Peritoneal adhesion. (1) peritoneal adhesions diagnosed by microlaparoscopy or abdominal operations, and classification according to Nair criteria is performed. (1) must be met. (2) Peritoneal adhesion symptoms, intermittent abdominal pain, abdominal distension, nausea and vomiting, hard to pass stools or gas; (3) Peritoneal adhesion signs，abdominal distension, abdominal tenderness, reduced or absent bowel sounds; (4) B ultrasound or CT or MRI show peritoneal adhesion or adhesion-related complications.

Exclusion Criteria:

1. Complete intestinal obstruction and suitable for surgery.
2. Patients known to be allergic to bevacizumab or any of the components of the drug.
3. Other ongoing anti-tumor treatment.
4. Heart disease with significant clinical symptoms, such as: congestive heart failure, coronary heart disease with symptom, arrhythmia hardly be controlled by drugs, myocardial infarction in 6 months, or heart failure
5. Active wound infection and a history of uncontrolled psychiatric illness.

   -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal adhesion ORR (pORR) | 3weeks after the last treatment
  Degree of adhesion was measured according to NAIR's criteria by laparoscopy. Grade 0 corresponded to no adhesions, Grade 1 and 2 corresponded to filmy adhesions and grade 3 and 4 to dense adhesions. No adhesions is defined as CR, dense adhesions change to filmy adhesions is defined as PR. The total efficiency ORR was calculated by taking the sum of CR+PR.

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | From first dose up to 1 month after the last treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Quality of Life (QoL) | From first dose up to 1 year
  Quality of Life (QoL) assessed by FACT-O
Progression free survival (PFS) | Up to 3 years
  From randomization until documented progressive disease or death
Overall survival (OS) | Up to 3 years
  From randomization until death
Objective Response Rate (ORR) | Up to 1 year
  The proportion of patients that have a best overall response of complete response (CR) or partial response (PR), as assessed by RECIST 1.1.

OTHER OUTCOMES:
Expression of VEGF-A in peritoneal cavity | Up to 1 year
  Quantitation of VEGF-A by enzyme-linked immunosorbent assay (ELISA), before and after intraperitoneal administration.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Du, PhD, Study Director — PLA 304 hospital
Locations (1):
- First Affiliated Hospital, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961